CLINICAL TRIAL: NCT04539366
Title: GD2-CAR PERSIST: Production and Engineering of GD2-Targeted, Receptor Modified T Cells (GD2CART) for Osteosarcoma or Neuroblastoma to Increase Systemic Tumor Exposure
Brief Title: Testing a New Immune Cell Therapy, GD2-Targeted Modified T-cells (GD2CART), in Children, Adolescents, and Young Adults With Relapsed/Refractory Osteosarcoma and Neuroblastoma, The GD2-CAR PERSIST Trial
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - review of safety data
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06646; NCI-2020-06646 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PED-CITN-02 (Other: Pediatric Early Phase Clinical Trial Network); PED-CITN-02 (Other: CTEP); U24CA224309 (NIH); UM1CA154967 (NIH); UM1CA228823 (NIH)
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Childhood Neuroblastoma; Recurrent Childhood Osteosarcoma; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Refractory Childhood Neuroblastoma; Refractory Childhood Osteosarcoma; Refractory Neuroblastoma; Refractory Osteosarcoma
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma | interventions — Biopsy; Specimen Handling; Cyclophosphamide; fludarabine phosphate; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (GD2 CAR T) (Experimental): LYMPHODEPLETION CHEMOTHERAPY: Patients receive fludarabine phosphate IV daily on days -5 to -2 and cyclophosphamide IV daily on days -4 to -2.
  GD2CART: Patients receive GD2CART cells IV on day 0.
  Patients also undergo ECHO, MUGA or cardiac MRI scan during screening, blood sample collection throughout the trial, and tumor biopsies and bone marrow aspiration and biopsy as clinically indicated. In addition, patients undergo standard imaging scans throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine Phosphate; Biological: GD2-CAR-expressing Autologous T-lymphocytes; Procedure: Imaging Procedure; Procedure: Magnetic Resonance Imaging of the Heart; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: GD2-CAR-expressing Autologous T-lymphocytes — Given IV
  Other Names: tvs-CTL Vaccine
Procedure: Imaging Procedure — Undergo standard imaging scans
  Other Names: Diagnostic Imaging Technique; Image Type; Imaging; Imaging (procedure); Imaging Procedures; Imaging Technique; imaging type; IMAGING_METHOD; imaging_type; Medical Imaging; Type of imaging
Procedure: Magnetic Resonance Imaging of the Heart — Undergo cardiac MRI
  Other Names: Cardiac MRI; Heart MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial investigates the side effects and determines the best dose of an immune cell therapy called GD2CART, as well as how well it works in treating patients with osteosarcoma or neuroblastoma that has come back (relapsed) or does not respond to treatment (refractory). T cells are infection fighting blood cells that can kill tumor cells. The T cells given in this trial will come from the patient and will have a new gene put in them that makes them able to recognize GD2, a protein on the surface of tumor cells. These GD2-specific T cells may help the body's immune system identify and kill GD2 positive tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of producing T cells modified to express a GD2-specific chimeric antigen receptor (GD2-CAR-expressing autologous T-lymphocytes [GD2CART]) meeting established release criteria using a dasatinib containing culture platform and retroviral vector in the Miltenyi CliniMACS Prodigy (Registered Trademark) system.

II. Determine the safety and maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) via administration of escalating doses of autologous GD2CART in children and young adults with relapsed/refractory osteosarcoma and neuroblastoma following cyclophosphamide-fludarabine based lymphodepletion.

III. Determine clinical activity in a preliminary fashion of autologous GD2CART in children and young adults with relapsed, refractory osteosarcoma and neuroblastoma.

SECONDARY OBJECTIVES:

I. Measure persistence of adoptively transferred GD2CART and correlate this with antitumor effects.

II. If unacceptable toxicity occurs that is possibly, probably, or definitely related to GD2CART, assess the capacity for rimiducid (AP1903), a dimerizing agent, to mediate clearance of the genetically engineered cells and resolve toxicity.

III. Describe the feasibility and tolerability of a second infusion of GD2CART in select patients.

EXPLORATORY OBJECTIVES:

I. Compare persistence of GD2CART administered in this trial to that observed in a previous trial using GD2.OX40.28.z.iCasp9 CAR T cells (NCI 14-C-0059) and assess features of the T cell product and the expanded T cells in vivo that correlate with persistence.

II. Conduct exploratory studies measuring levels of circulating myeloid cells including myeloid derived suppressor cells (MDSCs) in patients treated on this trial and compare levels to those observed in NCI 14-C-0059.

III. Explore GD2 expression in patients with neuroblastoma and osteosarcoma, including patients who have previously received anti-GD2 antibodies, from tissue and/or bone marrow samples at study entry and if available, after cell infusion.

OUTLINE: This is a dose-escalation study of GD2CART followed by a dose-expansion study.

LYMPHODEPLETION CHEMOTHERAPY: Patients receive fludarabine phosphate intravenously (IV) daily on days -5 to -2 and cyclophosphamide IV daily on days -4 to -2.

GD2CART: Patients receive GD2CART cells IV on day 0.

Patients also undergo echocardiogram (ECHO), multigated acquisition scan (MUGA) or cardiac magnetic resonance imaging (MRI) scan during screening, blood sample collection throughout the trial, and tumor biopsies and bone marrow aspiration and biopsy as clinically indicated. In addition, patients undergo standard imaging scans throughout the trial.

After completion of study treatment, patients are followed up three times weekly until day 14, twice weekly until day 28, at months 2, 3, 6, 9, and 12, every 3 months until the end of the second year, then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed neuroblastoma or osteosarcoma that is recurrent or refractory and for which standard curative measures do not exist or are no longer effective. Must have histologic verification of their disease at diagnosis or at relapse
* Patients with osteosarcoma in the dose escalation cohort, must have evaluable or measurable disease at enrollment
* Patients with osteosarcoma in the expansion cohort must have measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) at enrollment
* Patients with neuroblastoma in the dose escalation or dose the expansion cohort must have:

  * Prior progressive disease OR refractory disease present since diagnosis AND at least one of the following:

    * Evidence of tumor in the bone marrow (BM)
    * At least one metaiodobenzylguanidine (MIBG)-avid soft tissue or skeletal site
    * For MIBG-nonavid disease, at least one FDG-PET- positive soft tissue or skeletal site plus past histologic confirmation
  * Progressive disease is defined as any disease progression occurring at any time after the diagnosis of high-risk neuroblastoma. Refractory disease is defined as an incomplete response of high-risk neuroblastoma to all treatments but without disease progression
* Must be < 40 years of age
* There is no limit to the number of prior treatment regimens. The following washout periods prior to leukapheresis apply to patients undergoing leukapheresis on this study. If a patient has cryopreserved peripheral blood mononuclear cells (PBMCs) stored, the following washout periods are strongly recommended but not required and the product is useable if it meets the criteria established in this Investigational New Drug (IND)

  * Myelosuppressive chemotherapy: Patients must not have received myelosuppressive chemotherapy within 3 weeks of leukapheresis (6 weeks if prior nitrosourea)
  * Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a short-acting growth factor. At least 14 days must have elapsed after receiving pegfilgrastim
  * Biological agent, tyrosine kinase inhibitor, targeted agent, metronomic chemotherapy: At least 7 days must have elapsed since the completion of therapy with a biologic agent, tyrosine kinase inhibitor, targeted agent, or metronomic non-myelosuppressive regimen
  * 131I-MIBG or other radioisotope therapy: At least 6 weeks must have elapsed since prior therapy with 131I-MIBG. At least 6 weeks or 10 half-lives (whichever is shorter) must have elapsed since prior therapy with any other radioisotope
  * Monoclonal antibodies and checkpoint inhibitors: At least 3 weeks or 5 half-lives (whichever is shorter) must have elapsed since prior therapy that included a monoclonal antibody or checkpoint inhibitor
  * Radiotherapy (XRT): 3 weeks must have elapsed since XRT; at least 6 weeks if XRT involved central nervous system (CNS) or lung fields; and at least 12 weeks from total-body irradiation (TBI), craniospinal XRT, or XRT involving ≥ 50% bony pelvis, with the exception that there is no time restriction for palliative radiation with minimal bone marrow involvement and the patient has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression
  * Vaccine therapy, anti-GD2 mAb therapy, or therapy with any genetically engineered T cells: Patients may have received previous vaccine therapy, anti-GD2 monoclonal antibody (mAb) therapy, or therapy with any genetically engineered T cells except prior GD2 CAR T cell therapy. At least 3 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior vaccine or monoclonal antibody therapy. At least 42 days must have elapsed since prior modified T cell, natural killer (NK) cell, or dendritic cell therapy
  * Allogeneic stem cell transplant/infusion: At least 12 weeks must have elapsed since allogeneic stem cell transplant and without evidence of active graft versus host disease (GVHD)
  * Autologous stem cell transplant/infusion: Patients who received an autologous stem cell infusion following myeloablative therapy should be at least 6 weeks from their infusion. Patients who received an autologous stem cell infusion following non-myeloablative therapy do not have a wash-out period; they are eligible once they meet all other eligibility requirements, including recovery from acute side effects
* Must meet parameters for apheresis per institutional guidelines. (This criterion does not apply to patients with apheresis product or usable T cell product available for use). Cryopreserved PBMCs stored from participation in other institutional cell therapy or cell collection studies or standard of care may be used to generate the cellular product on this study if they meet the criteria established in this IND
* Patients > 16 years of age must have Karnofsky ≥ 60%. Patients ≤ 16 years of age must have Lansky scale ≥ 60%; corresponding to Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Leukocytes >= 750/mcL (For patients without bone marrow involvement. Patients who have bone marrow involvement with tumor are exempt from the platelet requirement and will not be evaluable for hematological toxicities. Patients must not be refractory to transfusions)
* Absolute neutrophil count (ANC) ≥ 500/mcL (For patients without bone marrow involvement. Patients who have bone marrow involvement with tumor are exempt from the platelet requirement and will not be evaluable for hematological toxicities. Patients must not be refractory to transfusions.)
* Platelets >= 75,000/mcL (transfusion independent defined as no transfusion in prior 7 days) (For patients without bone marrow involvement. Patients who have bone marrow involvement with tumor are exempt from the platelet requirement and will not be evaluable for hematological toxicities. Patients must not be refractory to transfusions.)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 5 x upper limit of normal (ULN) (For the purpose of this study, the ULN for SGOT is 50 U/L and the ULN for SGPT is 45 U/L)
* Albumin >= 2 g/dL
* Total bilirubin =< 2 x institutional upper limit of normal (ULN) for age. Patients with Gilbert's syndrome are excluded from the requirement of a normal bilirubin and patients will not be excluded if bilirubin elevation is due to tumor involvement. (Gilbert's syndrome is found in 3-10% of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis). Note: Adult values will be used for calculating hepatic toxicity and determining eligibility
* Age, maximum serum creatinine (mg/dL):

  * 1 month to < 6 months: 0.4 (male), 0.4 (female)
  * 6 months to < 1 year: 0.5 (male), 0.5 (female)
  * 1 to < 2 years: 0.6 (male), 0.6 (female)
  * 2 to < 6 years: 0.8 (male), 0.8 (female)
  * 6 to < 10 years: 1 (male), 1 (female)
  * 10 to < 13 years: 1.2 (male), 1.2 (female)
  * 13 to < 16 years: 1.5 (male), 1.2 (female)
  * >= 16 years: 1.7 (male), 1.4 (female) OR Creatinine clearance or glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 for patients with levels above institutional normal
* Cardiac ejection fraction >= 45% or shortening fraction >= 28%, no evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO). No clinically significant electrocardiogram (ECG) findings
* Pulmonary status: No clinically significant pleural effusion. Baseline oxygen saturation > 92% on room air at rest
* No acute neurotoxicity greater than grade 2 with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible
* Females of child-bearing potential and males of reproductive potential who are sexually active must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the start of study enrollment until 6 months after GD2 CAR T cell infusion (or until the duration of study participation, in the case of patients who start lymphodepleting chemotherapy but do not receive the GD2 CART infusion). Should a female become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * Note: Females of childbearing potential are defined as those who are past the onset of menarche and are not surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, complete hysterectomy) or post menopausal
* All patients >= 18 years of age must be able to give informed consent or if unable to give consent have a legal authorized representative (LAR) who can give consent for the patient. For patients < 18 years old their LAR (i.e., parent or legal guardian) must give informed consent. Pediatric patients will be included in age appropriate discussion and verbal assent will be obtained for those > 7 years of age, when appropriate, according to local policy

Exclusion Criteria:

* Receiving any other current investigational agents
* History of anaphylactic reactions attributed to anti-GD2 antibodies or to compounds of similar chemical or biologic composition to GD2CART, cyclophosphamide, fludarabine, or other agents used in this study. History of hypersensitivity to dornase alfa, Chinese hamster ovary cell products, or any of the components of pulmozyme
* Patients who require systemic corticosteroid or other immunosuppressive therapy. (A one-week washout from systemic corticosteroid or other immunosuppressive therapy is permitted.) Use of physiologic doses of corticosteroids (up to 3 mg/m^2/day prednisone equivalent) are permitted. Use of topical, ocular, intra-articular, intra-nasal, or inhaled corticosteroids are permitted
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of additional malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast) unless untreated and stable or disease free for at least 3 years
* Untreated central nervous system (CNS) metastasis. Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are permitted. Patients who are clinically stable as evidenced by no requirements for corticosteroids, no evolving neurologic deficits, and no progression of residual brain abnormalities without specific therapy, are permitted. Patients with asymptomatic subcentemeric CNS lesions are permitted if no immediate radiation or surgery is indicated
* CNS disorder such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or autoimmune disease with CNS involvement that in the judgement of the investigator may impair the ability to evaluate neurotoxicity
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled
* Ongoing infection with human immunodeficiency virus (HIV), hepatitis B (hepatitis B surface antigen [HBsAg] positive), or hepatitis C virus (anti-HCV positive) as the immunosuppression contained in this study will pose unacceptable risk. A history of HIV, hepatitis B, or hepatitis C is permitted if the viral load is undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing
* Primary immunodeficiency or history of systemic autoimmune disease (e.g., Crohns, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
* Females of childbearing potential must have a negative serum or urine pregnancy test. Pregnant females are excluded from this study because the effects of autologous GD2CART on the developing human fetus are unknown and because the chemotherapy agents used in this trial (cyclophosphamide and fludarabine) are category D agents with the potential for teratogenic or abortifacient effects. Additionally, because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with cyclophosphamide/fludarabine, breastfeeding should be discontinued if the mother is treated with cyclophosphamide/fludarabine. These potential risks may also apply to other agents used in this study
* In the investigator's judgment, unlikely to complete protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation. Or in the investigator's judgment, if the patient is likely to develop significant toxicity and morbidity from CAR-T cell expansion mediated inflammation based on location of tumor site

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of producing GD2-CAR-expressing autologous T-lymphocytes (GD2CART) cells | Up to day 28 days after cell infusion
  Success will be defined by manufacturing and expansion of GD2CART to satisfy the targeted dose level and meet the requirements of the Certificate of Analysis. Specifically, dose escalation will proceed if 3 or more of the first 3 to 6 patients in a dose level are able to produce adequate cells for evaluation.
Incidence of adverse events (AEs) | Up to 15 years
  Safety of GD2CART will be by the incidence and severity of dose limiting toxicities, treatment emergent AEs, serious adverse events, laboratory abnormalities, changes in vital signs, and changes in physical examination following infusion of GD2CART cells.
Maximum tolerated dose | Up to day 28 days after cell infusion
  Estimate of the maximum tolerated dose of autologous GD2CART in children and young adults with relapsed/refractory osteosarcoma and neuroblastoma following cyclophosphamide-fludarabine based lymphodepletion defined as the dose at which less than 33% of evaluable patients experience a cycle 1 dose limiting toxicity.
Best response to GD2CART cells | Up to day 28 days after cell infusion
  Simon's two stage design will be used to evaluate the clinical benefit of GD2CART after conditioning lymphodepletion chemotherapy in two groups of patients: children and young adults with recurrent, refractory osteosarcoma and neuroblastoma.

SECONDARY OUTCOMES:
Persistence of GD2CART cells | Up to 5 years
  Persistence of GD2CART and correlation with tumor regression and sustained clinical benefit will be assessed. Persistence will be defined as the duration of time that GD2CART cells can be detected above the background rate (baseline measure) as measured by polymerase chain reaction. The persistence will be compared between the different response statuses (responders versus non-responders) using a t-test allowing for unequal variance.
Capacity for rimiducid (AP1903) to reverse unacceptable toxicity related to GD2CART administration | Up to 28 days after cell infusion
  The toxicity is defined to be reversed or resolved when the toxicity grading has resolved to grade 2 or below. The resolution of toxicity will be summarized descriptively.
Feasibility and tolerability of a second infusion of GD2CART cells | After a 2nd infusion of GD2CART cells
  The proportion of evaluable patients who produce adequate GD2CART produced that meet Certificate of Analysis (COA) for infusion.

OTHER OUTCOMES:
Persistence of GD2CART cells | Up to 15 years
  Associations between biomarkers and chimeric antigen receptor persistence will be assessed by regression. The exact statistical model will depend on the observed responses which might not be linearly related to biomarkers but could show logistic or other association. Relationships of biomarkers to outcomes (overall survival, progression free survival) will be assessed by Cox regression using baseline measurements as predictors. The proportional hazards assumption will be checked retrospectively.
Biomarkers | Up to 28 days after cell infusion
  Will measure levels of circulating myeloid cells including myeloid derived suppressor cells in patients treated on this trial and compare levels to those observed in NCI 14-C-0059.
GD2 expression | Up to 28 days after cell infusion
  Tumor and/or normal tissue will be obtained from archival sample, tissue or tumor biopsy, or any clinically indicated surgeries. Bone marrow aspirations will be conducted in all patients with neuroblastoma. In patients with osteosarcoma, bone marrow aspirations will be conducted only if clinically indicated, i.e. known bone marrow involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Rosandra N Kaplan, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm